CLINICAL TRIAL: NCT05749354
Title: Clinical Study of Liver Meridian in the Treatment of Male Impotence and Female Premature Ovarian Failure
Brief Title: Clinical Efficacy of Acupuncture on the Liver Meridian in Men With Erectile Dysfunction Reserve
Acronym: GJZLBQGNZA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019YFC1709104
Record Dates: First submitted 2023-01-12; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Erectile Dysfunction; Acupuncture Therapy; Median Nerve Disease
MeSH Terms: conditions — Erectile Dysfunction; Median Neuropathy | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- liver meridian group (Experimental): Four acupoints; LR3 Taichong, LR5 Ligou, LR8 Ququan, and LR12 Jiman. Based on the national standard of the People's Republic of China in 2006 (GB/T 12346-2006). The patient will be in a supine position. Taichong will be punctured at a 25-mm depth using a 0.35×25-mm filiform needle, Ligou will be punctured at a 15-20-mm depth with a 0.35×25-mm filiform needle, Ququan at a 20-25-mm depth with a 0.30×40-mm filiform needle, and an acute pulse of 15-20 mm. Each acupoint will be subject to a small amount of uniform lifting and twisting to the degree of local acid distension. An auxiliary needle (0.16×13 mm) will be inserted approximately 5 mm into the needle, 2 mm proximal to the heart of each acupoint along the meridian. The negative electrode will be connected to the main point, and the positive electrode will be connected to the auxiliary needle, and connect the electroacupuncture instrument. The needles will be retained for 30 min respectively, once every other day, 24 treatments.
  Interventions: Other: electroacupuncture
- stomach meridian group (Active Comparator): Four acupoints have been selected for the gastric meridian group, including ST42 Chongyang, ST40 Fenglong, ST36 Zusanli, and ST31 Biguan. The acupoint locations are based on the national standard of the People's Republic of China in 2006 (GB/T 12346-2006). The patient will be supine during the procedure, and the needles will be routinely sterilized. Straight needling will be performed in the hip region using a 0.30×50-mm-filiform needle, a 0.30×50-mm filiform needle in Zusanli, and a 0.30×40-mm filiform needle in Fenglong. A 0.35×25-mm filiform needle will be used to stimulate Chongyang for 10-15 mm, and each acupoint will be gently and evenly lifted, inserted, and twisted to local acid distension. Electroacupuncture will be applied in the same manner as for the liver meridian group. The needles will be retained for 30 min respectively, once every other day, then thrice weekly for a total of 24 treatments in the three groups.
  Interventions: Other: electroacupuncture
- non-acupoint group (Placebo Comparator): Four points: (1) On the lateral thigh, between the vastus lateralis and biceps femoris, the midpoint of the popliteal stria, and the highest point of the greater trochanter. (2) On the lateral side of the calf, beside the level of Zusanli, and at the lateral edge of the tibia. (3) On the fibular side of the calf, the midpoint of the stomach meridian, and the bile meridian, 3 cm above the tip of the lateral malleolus and in front of the hanging bell. (4) On the lateral side of the calcaneus, and the servant enters the midpoint of the line connecting the posterior edge of the calcaneus at the same level. The 0.30×25-mm filiform needles are inserted straight for 3-5 mm at the points, the needles can stand without Deqi. The auxiliary needle will be inserted and electroacupuncture will be connected (same as in the other group). The internal wire of the electroacupuncture instrument will be interrupted, no current passed through. The treatment time is the same as the other two groups.
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — Electroacupuncture (EA) is a method of treating diseases by inserting a needle (usually a filiform needle) into the skin or tissue of a patient at a certain Angle, and then passing through the needle (sensing) micro-current waves of human bioelectricity to stimulate specific parts of the human body (acupoints).
  1. Disposable sterile acupuncture filiform needle (0.16mm×13mm, 0.30mm×25mm, 0.30mm× 40mm), Guizhou Andi Medical Equipment Co, LTD, Guizhou Food and Drug Supervision and Equipment Production Xu 20170011.
  2. Electroacupuncture apparatus: SDZ-Ⅱ electroacupuncture apparatus of Huatuo brand, Suzhou Medical Supplies Factory Co., LTD., Registration No. : 20172270675.
  For non-acupoint group,the internal wire of the electroacupuncture instrument will be interrupted, no current passed through.
  Other Names: acupuncture

SUMMARY:
Erectile dysfunction (ED) is a kind of worldwide and common sexual dysfunction disease, which mainly affects men over forty years old. The clinical characteristics of ED is the inability to maintain sufficient erection to obtain satisfactory sexual intercourse. Age, education, diabetes, stroke, obesity, and hypertension are factors inducing ED. Recent years, the prevalence of ED is rising, and more men aged below forty years old are suffering ED. Published review indicated that the prevalence of ED was 40.56% in Chinese men aged over forty years old. A survey conducted in China suggested that 40.56% men aged over forty years old suffered from ED. Another international survey found that, 21.48% sexually active participants suffered from ED. Several researches demonstrated that, ED affects health and quality of life of patients and partner. Besides, ED induces patients' psychosocial problems, including depression and anxiety, and reduce work efficiency. According to American Urological Association guideline published in 2018, the clinical therapies for ED include phosphodiesterase type 5 inhibitor (PDE5i), vacuum erection device, and penile prosthesis implantation. PDE5i (such as sildenafil, vardenafil, and tadalafil) is a first-line drug for ED, recommended by doctors and patients. However, the most common side effects of PDE5i were headache, dyspepsia, flushing, and blurred vision. Furthermore, the ideal dose and type of PDE5i still need to be further studied. The use of PDE5i is restricted by those reasons.

Acupuncture is an important role of Traditional Chinese Medicine (TCM), and acupuncture received more concerned recently. The correlation between meridians and viscera is the center of acupuncture scientific problem. Acupoints stimulation can regulate visceral sensation and mobility to treat diseases.

DETAILED DESCRIPTION:
This is a three-arm, multi-center, randomized controlled trial. Participants will be recruited in this study, with participants in each group. This trial is reported on the basis of the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines and complies with the principles of the Consolidated Standards of Reporting Trials (CONSORT) and Standards for Reporting Interventions in Clinical Trial of Acupuncture (STRICTA).The study will be carried out from January 2023 to December 2023 at five hospitals in China. Those hospitals include the first hospital of Hunan university of Chinese Medicine, Chengdu university of traditional Chinese medicine, Jiangsu Province Hospital of Chinese Medicine, The Affiliated Hospital of Jiangxi University of TCM, and Guizhou university of TCM. This research will recruit participants with ED by outpatient and inpatient department and social media. The patients who meet the diagnostic criteria of American Urological Association will be included in this study. The eligible patients with ED will be allocated into three groups: the liver meridian group, the stomach meridian group, and the non-acupoint group in a 1:1:1 ratio. The total observation period is twenty weeks, including a one-week baseline, eight-week treatment period, and twelve-week follow-up period. Outcome evaluation will be implemented at the baseline, during the treatment period, and during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 22 and 50 years
* Having a sexual partner and having regular sex life at least twice a week
* Meeting the diagnostic criteria of ED
* The scores of IIEF-5 between 8 points to 21 points
* PDE5i or similar medication weren't taken one month before treatment
* Patients agree to participate in this study.

Exclusion Criteria:

* Congenital genital malformation and dysplasia
* Severe reproductive system infection
* ED induced by genitourinary surgery and lower abdominal surgery
* Severe cardiovascular disease, liver disease, kidney disease
* Severe hypertension, diabetes, and blood diseases have not been controlled
* Severe mental illness
* Contraindications of PDE5i.

Ages: 22 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
5-item version of the International Index of Erectile Function (IIEF-5) | Baseline period,enrollment 2 weeks, enrollment 4 weeks, enrollment 6 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  In this trial, the 5-item version of IIEF will be applied as primary outcome. The IIEF-5 contains 5 questions and measures the erectile function and intercourse satisfaction. Responses are rated on 5-point Likert scales for every item. The total scores of all 5 items are the overall IIEF-5 score.

SECONDARY OUTCOMES:
Sexual Encounter Profile (SEP) diaries | Baseline period,enrollment 2 weeks, enrollment 4 weeks, enrollment 6 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  In this trial, the development of sexual activity will be assessed using the Sexual Encounter Profile (SEP) diaries (SEP-Questions 2 and 3). After each sexual intercourse, the participants will be asked to record the following two yes/no questions of the test: SEP Question 2: " Were you able to insert your penis into your partner's vagina?" SEP3 Question 3: " Did your erection last long enough for you to have successful intercourse? ".
Erectile hardness grading scale (EHS) | Baseline period,enrollment 2 weeks, enrollment 4 weeks, enrollment 6 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  To investigate the erectile hardness, the erectile hardness grading scale (EHS) was used in this trial. According to the EHS, the erectile hardness is divided into four grades. Grade one of EHS is that penis enlarged but not hard. Grade two of EHS is that the penis is slightly erect, but not enough for penetration. Grade three of EHS is that penis erection hard for penetration but not hard completely. Grade four of EHS is that penis is completely hard and fully rigid.
Treatment satisfaction scale (TSS) | Baseline period,enrollment 2 weeks, enrollment 4 weeks, enrollment 6 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  The treatment effectiveness for both patients and partners will be measured using The Treatment Satisfaction Scale (TSS) . The TSS questionnaire consist of four parts, including unmedicated patient, medicated patient, unmedicated partner, and medicated partner modules. The content of TSS include the satisfaction with sexual spontaneity, quality of erection, quality of ejaculation, sexual pleasure, orgasm, confidence, reliability of treatment, side effects, convenience, overall satisfaction, conformity to treatment expectations and intent to continue treatment.
The Hamilton Anxiety Scale (HAMA) | Baseline period, enrollment 4 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  The symptoms of anxiety induced by ED will be evaluated by The Hamilton Anxiety Scale (HAMA) separately. The higher the score, the heavier anxiety.
The Hamilton Depression Scale (HAMD) | Baseline period, enrollment 4 weeks, enrollment 8 weeks, enrollment 12 weeks, enrollment 16 weeks, enrollment 20 weeks（changes from Baseline at 8 weeks of treatment and 12 weeks of follow-up）
  The symptoms of depression induced by ED will be evaluated by The Hamilton Depression Scale (HAMD) separately. The higher the score, the heavier the depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Our subject database is called Zintuikang Integrated Big Data Application Platform, and other researchers can access it through the website. The administrator set up the account, and other researchers can log in by changing the password after registration. Their account has the authority to access the data and enter the CRF form.

REFERENCES:
- [Background] Rong P, Zhu B, Li Y, Gao X, Ben H, Li Y, Li L, He W, Liu R, Yu L. Mechanism of acupuncture regulating visceral sensation and mobility. Front Med. 2011 Jun;5(2):151-6. doi: 10.1007/s11684-011-0129-7. Epub 2011 Jun 22. PMID 21695619
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Araujo AB, Allen KR, Ni X, Rosen RC. Minimal clinically important differences in the vaginal insertion and successful intercourse items of the sexual encounter profile. J Sex Med. 2012 Jan;9(1):169-79. doi: 10.1111/j.1743-6109.2011.02506.x. Epub 2011 Oct 7. PMID 21981744
- [Background] Mulhall JP, Goldstein I, Bushmakin AG, Cappelleri JC, Hvidsten K. Validation of the erection hardness score. J Sex Med. 2007 Nov;4(6):1626-34. doi: 10.1111/j.1743-6109.2007.00600.x. Epub 2007 Sep 21. PMID 17888069
- [Background] Kubin M, Trudeau E, Gondek K, Seignobos E, Fugl-Meyer AR. Early conceptual and linguistic development of a patient and partner treatment satisfaction scale (TSS) for erectile dysfunction. Eur Urol. 2004 Dec;46(6):768-74; discussion 774-5. doi: 10.1016/j.eururo.2004.08.001. PMID 15548446
- [Background] Maier W, Buller R, Philipp M, Heuser I. The Hamilton Anxiety Scale: reliability, validity and sensitivity to change in anxiety and depressive disorders. J Affect Disord. 1988 Jan-Feb;14(1):61-8. doi: 10.1016/0165-0327(88)90072-9. PMID 2963053
- [Background] Gjerris A, Bech P, Bojholm S, Bolwig TG, Kramp P, Clemmesen L, Andersen J, Jensen E, Rafaelsen OJ. The Hamilton Anxiety Scale. Evaluation of homogeneity and inter-observer reliability in patients with depressive disorders. J Affect Disord. 1983 May;5(2):163-70. doi: 10.1016/0165-0327(83)90009-5. PMID 6222096